CLINICAL TRIAL: NCT05032469
Title: Effect of The Foot Reflexology Applied Before Chest Tube Removal on the Pain And Anxiety Level: A Randomized Controlled Trial
Brief Title: Foot Reflexology to Reduce Pain and Anxiety Before Chest Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Elif BUDAK ERTÜRK, Principal Investigator, Assistant Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24074710-38
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Chest Tube Removal; Heart; Surgery, Heart, Functional Disturbance as Result; Pain; Anxiety
Keywords: Anxiety; Cardiac surgery; Chest tubes; Nursing; Pain; Reflexology
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refloxology Intervention (Experimental): The first foot reflexology was applied to the intervention group for 30 min (20 min on the right foot, 10 min on the left foot) on the first postoperative day (24 h after the surgery). On the second postoperative day, 30 min of foot reflexology was applied to the patients who decided to chest tube removal (CTR). After the foot reflexology applied by the researcher, CTR was performed by the doctor within 10 min. Immediately after CTR, the patient's pain and anxiety level during CTR was measured. At the 15th minute after CTR, the pain and anxiety level of the patients was measured, their satisfaction with the reflexology application was measured. Then, the patients were asked to describe the pain and feelings and thoughts during CTR, 1 hr after CTR, pain level was measured, and they were asked to express their feelings and thoughts about the reflexology application.
  Interventions: Other: Reflexology
- Standart Care (No Intervention): Participants in the control group will receive standart postoperative care.

INTERVENTIONS:
Other: Reflexology — Reflexology is a method that creates nervous, hormonal and energetic effects in the body using pressure, rubbing and stretching applied with special hand and finger techniques to reflex points corresponding to all parts, organs and systems of the body in the ears, hands and feet
  Arms: Refloxology Intervention

SUMMARY:
In open heart surgeries, patients experience severe pain due to tissue trauma, damage to intercostal nerves, and muscle spasm due to pulling tubes from the mediastinal space and between the pleural leaves pull during chet tube removal (CTR). When acute pain is not relieved, the patient develops emotional, psychological (eg post-traumatic stress disorder) and physical problems (eg chronic pain) after surgery. Since this situation negatively affects the healing process, it increases the anxiety level of the patients and decreases the comfort level. Reflexology is one of the non-pharmacological methods used in the management of pain and anxiety after open heart surgery The aim of this randomized controlled study was to identify the effect of foot reflexology applied before chest tube removal process on pain and anxiety level. This study will be done a randomized-controlled trial to test the intervention.

DETAILED DESCRIPTION:
Background: Patients undergoing cardiovascular surgery suffer from anxiety and pain due to the chest tube removal (CTR).

Objective/Hypothesis: The aim of this randomized controlled study was to identify the effect of foot reflexology applied before chest tube removal process on pain and anxiety level.The following hypotheses (H) were tested in this study:

H1a : There was a difference between the reflexology group and the control group in terms of pain level during CTR.

H1b : There was a difference between the reflexology group and the control group in terms of anxiety level during CTR.

H1c : There was a difference between the reflexology group and the control group in terms of the difference between the pain level before CTR and during CTR.

H1d : There was a difference between the reflexology group and the control group in terms of the difference between the anxiety level before CTR and during CTR.

Study design: A randomized controlled trial. Method: The study sample who has gone through coronary artery bypass graft surgery was randomly assigned to reflexology or the control group (twenty- eight each in). The primary outcomes were pain, evaluated using a numeric pain-rating scale, and anxiety evaluated by the profile of mood states scale tension-anxiety subscale, both measured first (before and after reflexology) and second postoperative days (before the reflexology and immediately after chest tube removal, 15th minutes and 1 h).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years who have CABG surgery
* Having at least two chest tube catheters
* Having chest tubes removed together
* Volunteering to participate in the research

Exclusion Criteria:

* Patients with diagnosed with psychiatric illness
* Having orientation or confusion problems, complete vision or hearing loss, mental problems due to problems such as dementia, mental retardation, and language problems
* Having pacemaker, varicose veins in the ankles
* Having chronic pain
* Having femoral fracture and open wound on the sole of the foot
* Having acute infection and hyperthermia, thromboembolism, suspected deep vein thrombosis at the postoperatively

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale Change | 1st postoperative day change from baseline pain score at after intervention, 2nd postoperative day change from baseline pain score at during, 15th min,1h after chest tube removal
  Numeric Pain Rating Scale includes values ranging from 0 (no pain) - 10 (the worst pain)
Profile of Mood States Scale Tension-Anxiety Subscale Change | 1st postoperative day change from baseline pain score at after intervention, 2nd postoperative day change from baseline pain score at during, 15th min after chest tube removal
  Profile of Mood States Scale Tension-Anxiety Subscale includes the following nine items: tense, shaky, on edge, panicky, uneasy, restless, nervous and anxious. Each item was graded as 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a bit) or 4 (extremely) and the sum of the items is the total scale, varying from 0 (no tension-anxiety) - 36 (most tension-anxiety).

SECONDARY OUTCOMES:
Numerical Satisfaction Evaluation Form | Second postoperative day
  Numerical Satisfaction Evaluation Form includes values ranging from 0 (I am not satisfied), 10 (I am satisfied)
Form to determine the feelings and thoughts of the patients about reflexology application and chest tube removal | Second postoperative day
  Six open ended questions about the feelings and thoughts of the patients about reflexology application and chest tube removal.

CONTACTS AND LOCATIONS:
Overall Officials: Elif BUDAK ERTÜRK, MsN,RN, PhD, Principal Investigator — Başkent University, Faculty of Health Science, Department of Nursing
Locations (1):
- Baskent University Ankara Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No